CLINICAL TRIAL: NCT04104906
Title: Motor Control Training in Individuals With Subacromial Pain Syndrome: Randomized Controlled Trial
Brief Title: Motor Control Training in Individuals With Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSACO2019
Record Dates: First submitted 2019-06-28; First posted 2019-09-26 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Shoulder Pain
Keywords: Shoulder rehabilitation; Electromyography; Posture analysis
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- motor control training (Experimental): 8-week exercise program, twice a week, with motor control training
  Interventions: Other: motor control training
- exercises (Active Comparator): 8-week exercise program, twice a week.
  Interventions: Other: The exercise group

INTERVENTIONS:
Other: motor control training — The volunteers of the motor control group will initiate the exercises on a stable and rigid basis. These will be progressed with adding an unstable base as the volunteer gains motor learning (between the fourth and fifth week of the protocol). For the motor control group, two sets of 10 repetitions will be performed keeping in isometry for ten seconds each repetition.
  Arms: motor control training
Other: The exercise group — the protocol of strengthening and will have five elastic bands with different resistances available (extra-light, light, moderate, strong and extra-strong) for elbow flexion exercises progression, medial rotation and lateral rotation of the shoulder and scapular retraction.
  Arms: exercises

SUMMARY:
The porpusose of this study is to evaluate the repercussions of a motor control exercise protocol in patients with subacromial pain syndrome without indication of surgical repair.

DETAILED DESCRIPTION:
Methods: This is a randomized controlled trial which will be composed of volunteers of both genders, aged between 35 and 60 years. All volunteers will undergo pre-assessment (Av1): pain sensation, pain and function, shoulder range of motion, muscle strength, electromyographic activity and kinematics of the shoulder complex. After the initial evaluation, the volunteers will be randomly divided into two groups to carry out the intervention: exercises (GE - conventional exercises with elastic band) and motor control (GCM - motor control training). The intervention protocol will last eight weeks. After four weeks, the second assessment (AV2), similar to AV1, will be performed and the global change perception questionnaire will be added. At the end of the intervention protocol, the third evaluation (AV3), similar to AV2, will be performed. A follow-up will be performed after 4 weeks of the end of the intervention protocol, with the assessment being equal to AV3.

The project will be submitted to the Research Ethics Committee of the Federal University of Rio Grande do Norte through the national interface "Plataforma Brasil". The study will also be registered on the international clinical trial platform, ClinicalTrials.gov. The study will only begin after approval of the ethics and research committee. All volunteers should read and sign the terms of free and informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Present subacromial pain with a score greater than or equal to 2 (Visual Analog Scale) for more than 2 months;
* Positive Neer test;
* Positive Hawkins test;
* Positive Jobe test (pain);
* Positive Patte test (pain);
* Involvement of the supraspinatus and / or infraspinatus tendon (without degenerative characteristics) confirmed by Magnetic Nuclear Resonance (MRI) examination.

Exclusion Criteria:

* Intense pain during the evaluations;
* Fail to properly perform the evaluation procedures;
* Two consecutive or five alternating absences during the training protocol.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Shoulder pain | Change from baseline in shoulder pain at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Evaluation of pain level in the shoulder using the Numerical Pain Scale, graded from 0 to 10, where 0 indicates absence of pain and 10 indicates the worst pain imaginable.
Shoulder function | Change from baseline in shoulder function at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Evaluation of shoulder pain and function using the Disabilities of the Arm, Shoulder and Hand (DASH). The questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. The higher the score, the greater the functional disability.

SECONDARY OUTCOMES:
Root Mean Square (RMS) | Change from baseline in RMS at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Analyze of the electromyographic activity of the muscles shoulder complex, after 4 and 8 weeks of the protocol and a follow up of 4 weeks after the intervention protocol, by Root Mean Square (RMS)
The kinematics of the scapula | Change from baseline in kinematics of the scapular girdle at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Analyze the kinematics of the scapula and glenohumeral in the slow and habitual movements after 8 weeks of the protocol and a follow up of 4 weeks.
Peak of muscular torque | Change from baseline in peak of muscular torque at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Evaluate the peak of muscular torque, by means of the manual dynamometer 8 weeks of the protocol and a follow up of 4 weeks.
Peak torque time | Change from baseline in peak torque time at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Evaluate the peak torque time, using the manual dynamometer 8 weeks of the protocol and a follow up of 4 weeks.
Range of motion | Change from baseline in range of motion at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Measure the range of motion for flexion, hyperextension, internal and external shoulder rotation 8 weeks of protocol and a follow up of 4 weeks, through the inclinometer.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Jamilson S Brasileiro, Natal, Rio Grande do Norte
  - Karinna Sonálya Aires da Costa, Parnamirim, Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: No